CLINICAL TRIAL: NCT05899699
Title: Potential Combination Topical Therapy of Acne Vulgaris: a Randomized Controlled Trial Comparing Efficacy of DAP/FLU Micro-emulsion vs. Standard Therapy of Adapalene.
Brief Title: Effect of New Topical Preparation for Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amgad E Salem, pHD, Assistant lecturer, pharmaceutical department, faculty of pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A.S.2019-32
Record Dates: First submitted 2023-06-03; First posted 2023-06-12 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAP/FLU ME (Experimental): Acne vulgaris patients treated with the optimized topical combination ME contain DAP-FLU.
  Interventions: Drug: DAP-FLU ME
- Adapalene .1% gel (Active Comparator): Acne vulgaris patients treated with standard therapy of Adapalene.
  Interventions: Drug: Adapalene .1% gel

INTERVENTIONS:
Drug: DAP-FLU ME — Combination therapy of topical anti-inflammatory agent (Dapsone 5%) and anti-androgenic agent (Flutamide 2.5%) with anti-bacterial agent of micro-emulsion component (tea tree oil 5%)
  Arms: DAP/FLU ME
Drug: Adapalene .1% gel — Adapalene .1% gel
  Arms: Adapalene .1% gel

SUMMARY:
The investigators propose a randomized, double-blind control trial study to evaluate the efficacy and safety of the optimized topical combination ME of the investigated drugs in the treatment of acne vulgaris containing DAP-FLU in comparison with standard therapy of Adapalene at Mansoura University Dermatology and Andrology Outpatient Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females age 12 or older
2. Clinical diagnosis of mild to moderate facial acne vulgaris defined as:

   1. ≥ 5 inflammatory lesions, and;
   2. ≥ 10 non-inflammatory lesions, and;
   3. IGA 2-3
3. Willing to refrain from using any treatments, other than the investigational product, for acne present on the face. This includes the use of antibiotics for the treatment of acne.
4. Willing and able to provide informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Women were excluded if they were pregnant, nursing, or planning a pregnancy as were men with facial hair that would interfere with the assessments.
2. Continuous or planned use of tanning booths or excessive sun exposure, in the opinion of the Investigator.
3. Treatment with systemic corticosteroids within 28 days prior to baseline.
4. Two or more active nodular lesions.
5. Use of androgen receptor blockers (such as spironolactone or flutamide) in the 7 days prior to randomization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Michaelson's acne severity index (ASI) | 8 Weeks
  It's evaluated by counting non-inflammatory lesions (open and closed comedones) and inflammatory lesions (papules, pustules and nodules of at least 5 mm in diameter), and calculated as follows:
  ASI = (comedones x 0.5) + (papules x 1) + (pustules x 2) + (nodules x 3).
Safety assessment by the recording of patient-reported adverse events | 8 Weeks
  Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Amgad El-Sayed Salem, Study Director — Mansoura University; Elham A. Mohamed, Study Director — Mansoura University; Noha M. Saleh, Study Director — Mansoura University; Marwa Z. Mubarak, Study Director — Mansoura University; Galal M. Abdelghania, Principal Investigator — Mansoura University
Locations (1):
- Amgad El-Sayed Salem, Al Mansurah, Egypt